CLINICAL TRIAL: NCT07045636
Title: Microbial Modulation by PEMF on Paque Induced Mucositis in Dental Implants Placed in Human Jaws: Microbiome and Proteomic Analysis.
Brief Title: Microbiome Modulation by PEMF on Plaque Induced Mucositis in Human Jaws
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jamil awad shibli (Other)
Collaborators: Harvard School of Dental Medicine (Other); Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor-Investigator, Jamil awad shibli, Professor, University of Guarulhos
Organization: University of Guarulhos (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PEMF and mucositis
Record Dates: First submitted 2025-05-15; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Microbial Colonization; Peri-Implantitis
Keywords: dental implants; peri-implantitis; mucositis; microbiome; proteomic
MeSH Terms: conditions — Communicable Diseases; Peri-Implantitis; Mucositis

STUDY DESIGN:
Intervention Model Description: Control group (healing cap without PEMF); test group with PEMF Comparison with teeth x implants (with or without PEMF)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization and placebo MED (medical device not activated or activated for the PEMF)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEMF x Control (without PEMF) (Experimental): Test group - Activated MED (with PEMF) installed on the test implants during the 21 days
  Control group - Non-activated MED (without PEMF) installed and NOT activated on the control implants during 21 days
  Interventions: Other: PEMF abd Sham (control); Diagnostic Test: Teeth wih gingivits
- Dental implants x teeth (No Intervention): Comparison between tooth and implants (with and without PEMF)

INTERVENTIONS:
Other: PEMF abd Sham (control) — Dental implants receive MED that could (test) or could not (control/SHAM) be activated to emit PEMF
  Arms: PEMF x Control (without PEMF)
Diagnostic Test: Teeth wih gingivits — Comparison with dental implants
  Arms: PEMF x Control (without PEMF)

SUMMARY:
To evaluate the impact of Pulsed Electromagnetic Field (PEMF) on mucositis induced in humans around dental implants and correlate these possible effects with the proteomic profile of implants with and without PEMF and teeth. The hypothesis is that PEMF may modulate bacterial biofilm formation around dental implants and enhance the host response following plaque-induced peri-implant mucositis.

DETAILED DESCRIPTION:
As in natural teeth, bacterial colonization of the implant surface can trigger a reversible inflammatory process in the peri-implant soft tissue-defined mucositis. However, differences in the organization of peri-implant tissues may combat the progression of lesions associated with bacterial biofilm, resulting in a broader inflammatory infiltrate compared to periodontal tissues. Some previous studies have used electromagnetic pulses (PEMF-pulse electromagnetic fields) to modulate bacterial biofilm. Thus, the objective of this study will be to evaluate the host response pattern (proteomics, microbiome, and clinical) during the induction and progression of experimental gingivitis and mucositis in humans with the action of the electromagnetic pulse. Forty systemically healthy individuals will be included, who must present the need for two implant-supported restorations adjacent to the teeth. Individuals will receive oral hygiene instruction and professional prophylaxis fortnightly, 30 days before implant installation. The implants will be installed in time -60 days. After 60 days, at baseline, the healing abutment will be installed on the two implants, one conventional and the other with an electromagnetic pulse. At the same time, everyone will receive acetate plates to protect the selected areas (tooth and implants) during brushing, to be used for 21 days. Clinical periodontal parameters, microbiological (supragingival and subgingival biofilm), and immunological (crevicular fluid) collections will be obtained at 0, 3, 7, 14, 21, 42, and 60 days. The results will be evaluated for normality using the D'Agostino test. Then, parametric or non-parametric tests will be applied to compare the means/medians obtained between the gingivitis and mucositis groups in the different periods of the study.

ELIGIBILITY:
Inclusion Criteria: -healthy individuals over 18 years of age

* have at least 2 contiguous edentulous spaces
* more than 15 teeth
* have not undergone periodontal treatment for at least 6 months before the start of the study

Exclusion Criteria: - Individuals with extensive dental restorations;

* with periodontal disease stages II to IV
* with peri-implantitis and/or mucositis (Shibli et al. 2015);
* individuals requiring previous grafting for implant insertion;
* diabetics;
* smokers or former smokers;
* pregnant women; lactating women;
* use of antibiotics or oral antiseptics in the last 6 months .

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2025-05-11 (Actual); Primary Completion 2025-05-11 (Actual); Study Completion 2025-05-11 (Actual)

PRIMARY OUTCOMES:
Number of clusters of microorganism | time points 0, 3, 6, 7, 14, 21, 28, 42, and 60 days
  amount of genera and microbial species detected and/or altered (reduction and increase)

CONTACTS AND LOCATIONS:
Overall Officials: Jamil A Shibli, PhD, Principal Investigator — Guarulhos University; Cinthya Massari, DDS, Study Director — Guarulhos University
Locations (1):
- Guarulhos University, Guarulhos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Souza JGS, Azevedo F, Borges MHR, Costa RC, Shiba T, Barak S, Mayer Y, Figueiredo LC, Feres M, Barao VAR, Shibli JA. Microbiome modulation of implant-related infection by a novel miniaturized pulsed electromagnetic field device. NPJ Biofilms Microbiomes. 2025 Feb 26;11(1):36. doi: 10.1038/s41522-025-00667-0. PMID 40011461
- [Background] Parize G, Luana Jimenez G, Shibli JA, Siroma R, Caetano MW, Kim YJ, Braz-Silva PH, da Silva Martinho H, Pallos D. Evaluation of Peri-Implantitis through Fourier-Transform Infrared Spectroscopy on Saliva. J Proteome Res. 2025 Feb 7;24(2):639-648. doi: 10.1021/acs.jproteome.4c00707. Epub 2025 Jan 10. PMID 39792796
- [Background] Mayer Y, Shibli JA, Saada HA, Melo M, Gabay E, Barak S, Ginesin O. Pulsed Electromagnetic Therapy: Literature Review and Current Update. Braz Dent J. 2024 Oct 25;35:e246109. doi: 10.1590/0103-6440202406109. eCollection 2024. PMID 39476109
- [Background] Mayer Y, Khoury J, Horwitz J, Ginesin O, Canullo L, Gabay E, Giladi HZ. A novel nonsurgical therapy for peri-implantitis using focused pulsed electromagnetic field: A pilot randomized double-blind controlled clinical trial. Bioelectromagnetics. 2023 Oct-Dec;44(7-8):144-155. doi: 10.1002/bem.22481. Epub 2023 Sep 1. PMID 37655846
- [Background] Faveri M, Miquelleto DEC, Bueno-Silva B, Pingueiro JMS, Figueiredo LC, Dolkart O, Yakobson E, Barak S, Feres M, Shibli JA. Antimicrobial effects of a pulsed electromagnetic field: an in vitro polymicrobial periodontal subgingival biofilm model. Biofouling. 2020 Aug;36(7):862-869. doi: 10.1080/08927014.2020.1825694. Epub 2020 Sep 29. PMID 32993357

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-22): https://cdn.clinicaltrials.gov/large-docs/36/NCT07045636/Prot_SAP_000.pdf
  • Informed Consent Form (2023-11-22): https://cdn.clinicaltrials.gov/large-docs/36/NCT07045636/ICF_001.pdf